CLINICAL TRIAL: NCT04453683
Title: Airway Management in Morbidly Obese Patients: A Comparison of Intubating Laryngeal Mask Fastrack and Air Q as a Conduit for Fiberoptic Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba Mohamed EL -Asser,MD, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Intubation in morbid obese
Record Dates: First submitted 2020-06-28; First posted 2020-07-01 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Intubation; Difficult or Failed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I ( Air Q) (Active Comparator): nsertion of proper size Air-Q. ILA
  Interventions: Device: Air-Q. ILA insertion of proper size
- Group II (ILMA) (Active Comparator): nsertion of proper size ILMA
  Interventions: Device: ILMA insertion of proper size

INTERVENTIONS:
Device: Air-Q. ILA insertion of proper size — Success of fiberoptic guided intubation throuhgh Air Q supraglottic airway device
  Arms: Group I ( Air Q)
Device: ILMA insertion of proper size — Success of fiberoptic guided intubation throuhgh ILMA supraglottic airway device
  Arms: Group II (ILMA)

SUMMARY:
To compare air Q versus ILMA intubation in obese adult paralyzed patient

DETAILED DESCRIPTION:
Evaluate the process of endo-tracheal intubation through Air Q compared to through ILMA regarding number and duration of attempts, laryngeal view grade, time to removal of device over tube without dislodgement and any complication

ELIGIBILITY:
Inclusion Criteria:All morbidly obese patient defined as BMI >40 kg/m2 scheduled for an elective surgery requiring general anesthesia with tracheal intubation were enrolled on the day of their surgery.

ASA physical status (I-II)

Exclusion Criteria physical status of IV or V or had a history of impossible tracheal intubation or awake fibreoptic intubation or if preoperative evaluation showed limited mouth aperture <3.5 cm or showed evidence that an awake fiberoptic intubation or rapid sequence induction would be required patients at increased risk for aspiration of gastric contents, coagulopathy or those with unstable cervical spines or requiring nasal route for tracheal intubation

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
success rate of tracheal intubation through each device. | Within a maximum of 5 minutes to confirm success of tracheal intubation through each supraglottic airway devices
  success rate of tracheal intubation through each device is defined as end tidal carbon dioxide confirmed placement of TT within a maximum of 5 min tracheal intubation time

SECONDARY OUTCOMES:
Insertion time of supraglottic airway devices | It is about 13-19 second for insertion of supraglottic airway devices
  Time necessary for insertion was measured from the time the face mask was taken away until the appearance of Co2 on the capnograph while supraglottic airway device in place

CONTACTS AND LOCATIONS:
Overall Officials: Heba M EL-Asser, MD, Principal Investigator — Zagazig University; Khadiga M El Hossiney, MD, Study Chair — Zagazig University; Amani A Aly, Study Chair — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frappier J, Guenoun T, Journois D, Philippe H, Aka E, Cadi P, Silleran-Chassany J, Safran D. Airway management using the intubating laryngeal mask airway for the morbidly obese patient. Anesth Analg. 2003 May;96(5):1510-1515. doi: 10.1213/01.ANE.0000057003.91393.3C. PMID 12707159
- [Background] Karim YM, Swanson DE. Comparison of blind tracheal intubation through the intubating laryngeal mask airway (LMA Fastrach) and the Air-Q. Anaesthesia. 2011 Mar;66(3):185-90. doi: 10.1111/j.1365-2044.2011.06625.x. PMID 21320087